CLINICAL TRIAL: NCT03017313
Title: A Prospective Post Marketing Non Interventional Study to Evaluate the Criteria on Which Renewal of LHRH Analogue Treatment is Made in Patients With Prostate Cancer Locally Advanced or Metastatic.
Brief Title: To Evaluate the Criteria for Renewal of Luteinizing Hormone-Releasing Hormone (LHRH) Analogue Treatment in Prostate Cancer Patients
Acronym: ANAREN
Status: Completed | Type: Observational
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Other Study IDs: A-ES-52014-224
Record Dates: First submitted 2016-12-30; First posted 2017-01-11 (Estimated); Last update posted 2021-06-24 (Actual); Status verified 2021-06

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: LHRH analogues — 3-or 6-month formulations

SUMMARY:
The purpose of the study, is to determine the percentage of patients for whom the initial LHRH prescription has been renewed

ELIGIBILITY:
Inclusion Criteria:

* Adult men diagnosed of locally advanced or metastatic prostate cancer scheduled to receive androgen deprivation therapy with a 3 or 6 month LHRH analogue including those requiring neo-adjuvant or adjuvant androgen deprivation therapy in association with radiotherapy
* Patients having provided written informed consent
* Patients mentally fit for completing a self-administrated questionnaire

Exclusion Criteria:

* Patients participating in another clinical study at the time of inclusion
* Patients with another severe malignant disease
* Life expectancy of less than 12 months
* Patients already treated with a LHRH analogue within the last year

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Prostate cancer locally advanced or metastatic
Sampling Method: Non-Probability Sample
Enrollment: 510 (Actual)
Dates: Start 2017-07-13 (Actual); Primary Completion 2021-06-14 (Actual); Study Completion 2021-06-14 (Actual)

PRIMARY OUTCOMES:
Percentage of patients for whom the initial LHRH prescription (the prescription at the baseline visit) has been renewed at first follow-up visit (same type, same formulation). | First follow-up visit (occurs 3 to 6 months from baseline)

SECONDARY OUTCOMES:
Percentage of patients for whom the initial LHRH prescription has been renewed at each visit. | Baseline, between 3 to 6 months, 12 months, 18 months and 24 months
Percentage of patients having switched from a 3 months to a 6 months and also 6 months to 3 months formulation at each visit. | Baseline, between 3 to 6 months, 12 months, 18 months and 24 months
Percentage of patients starting a 6-month formulation at baseline. | Baseline
  The decision to prescribe a LHRH analogue as a 3- or 6-months formulation will be made prior to and independently from the decision to enroll the subject. This decision should be made in accordance with the usual medical practice of the concerned investigator.
Reasons leading to a switch from a 3 months to a 6 months formulation (patient) presented as proportion of patients | Baseline, between 3 to 6 months, 12 months, 18 months and 24 months
Reasons leading to a switch from a 3 months to a 6 months formulation (physician) presented as proportion of physicians | Baseline, between 3 to 6 months, 12 months, 18 months and 24 months
Criteria for choice of formulation at start of hormonal treatment taking into consideration the patient characteristics and his disease status. | Baseline
Change of the Quality of Life Questionnaire QLQ-PR25 score compared to baseline and each visit. | Baseline, between 3 to 6 months, 12 months, 18 months and 24 months
Correlation between physician and patient satisfaction and the evolution of the biological parameters (Prostate-specific antigen) | Baseline, between 3 to 6 months, 12 months, 18 months and 24 months
Percentage of patients for which the initial prescription (the prescription at the baseline visit) of a LHRH analogue (3 or 6 months) has been stopped and later on renewed (intermittent treatment) | Baseline, between 3 to 6 months, 12 months, 18 months and 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (27):
- Spain (27):
  - Hospital A Coruña, A Coruña
  - Hospital del Sureste, Arganda
  - Hospital San Agustín, Avilés
  - Hospital de Txagorritxu, Barakaldo
  - Hospital de Basurto, Bilbao
  - Hospital Gral. Univ. Santa Lucía, Cartagena
  - Hospital Arquitecto Marcide, Ferrol
  - Hospital Univ. de Getafe, Getafe
  - Hospital de Cabueñes, Gijón
  - Hospital Universitario Dr Negrín, Las Palmas de Gran Canaria
  - Hospital de León, León
  - Hospital de la Princesa, Madrid
  - Hospital Univ. La Paz, Madrid
  - Hospital Univ. Infanta Sofía, Madrid
  - Hospital de Torrejón, Madrid
  - Hospital Rey Juan Carlos, Madrid
  - Hospital Comarcal Santiago Apóstol, Miranda de Ebro
  - Hospital Uni. Virgen de la Arrixaca, Murcia
  - Hospital Ntra. Señora del Cristal, Ourense
  - Hospital Son Llàtzer, Palma
  - Hospital Virgen del Camino, Pamplona
  - Hospital de Montecelo, Pontevedra
  - Hospital Univ. de Salamanca, Salamanca
  - Hospital Universitario de Canarias, Santa Cruz de Tenerife
  - Hospital Clínico de Santiago, Santiago de Compostela
  - Hospital Clínico de Valladolid, Valladolid
  - Hospital Álvaro Cunqueiro, Vigo